CLINICAL TRIAL: NCT05843019
Title: Adherence in Global Airways - the Relationship Between Steroid Intake and the Impact on the Endocrine Axis, Bone Density, and Structure in Patients With Chronic Sinusitis and Asthma
Brief Title: Adherence in Global Airways - Steroid Intake and Effects on Chronic Rhinosinosinutis
Acronym: AGAS 2023
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Christiane Haase (Other)
Responsible Party: Sponsor-Investigator, Christiane Haase, Clinical nurse specialist and Phd-student, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: 2022-ENT-steroids
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Chronic Rhinosinusitis Without Nasal Polyps; Asthma; Chronic Rhinosinusitis With Nasal Polyps; Steroid-Induced Osteopenia (Diagnosis); Steroid-Induced Diabetes; Steroid-Induced Hyperglycemia
Keywords: Adherence; Nurse; Global airways; Steroids
MeSH Terms: conditions — Asthma; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cross sectional: The patients in the cross sectional study will have done a synactenstest to investigate how their own product of kortisol os after longterm use of systemic steroids.
  The group consists of patients referred to the Respiratory Clinic, ENT, RH, for evaluation of CRS/CRSwNP/CRSnNP and with or without asthma for biological treatment. They are classified according to the type of inflammation they have (type-2 or non-type-2), whether they have CRSwNP or CRSsNP, their adherence, comorbidity with asthma, and finally the severity of the disease. All patients are given standard questionnaires to assess CRS/CRSwNP/CRSnNP and asthma (STARR-15, SNOT22, ACQ, ACT, MARS-5-L/N, Fosterscore - routine questionnaires for all patients in the Respiratory Clinic).

SUMMARY:
The purpose of this study is to investigate the relationship between long-term use of systemic steroids in patients with upper and lower respiratory tract diseases and their own production of cortisol (cross-sectional), as well as whether those with low cortisol levels have an impact on bone density. As patients with CRSwNP have a high use of steroids, they routinely undergo a DEXA scan at the Respiratory Clinic, Department of Ear-Nose-Throat Surgery and Audiology (ENT) - Rigshospitalet (RH) to examine whether their bone density and structure are affected. The scan will be included as a clinical secondary outcome to assess whether systemic steroid use has an impact on this.

The purpose of the study is therefore to compare steroid intake, baseline P-cortisol, the body's response to ACTH (measured by cortisol levels after the test), and bone density in patients with chronic sinusitis (CRS) with and without asthma in an unselected population at the Respiratory Clinic (cross-sectional). In addition, at the 4-month follow-up (exploratory follow-up, pilot project), it will be investigated whether good adherence (>80%) to inhalation therapy (nasal steroid and lung steroid) and additional treatment with biologicals has a negative effect on the body's own production of P-cortisol.

ELIGIBILITY:
Inclusion Criteria: cross sectional study

* Diagnosed with chronic rhinosinusitis (CRS)
* possibly asthma
* Aged over 18 years

Exclusion Criteria - cross sectional study

* Unable to read or speak Danish
* Presence of severe psychiatric comorbidities
* Patients who have never taken systemic steroids
* Inability to participate or comply with local treatment according to the investigators' assessment
* Does not provide consent for lookup in FMK-online

In/exclusion criteria for exploratory study - 4-month follow-up (pilot project)

Inclusion criteria:

* Diagnosed with CRS and possibly asthma
* Age over 18 years
* Low adherence: Foster score, i.e. the number of treatments taken compared to prescribed < 80% (4 weeks out of 16 weeks) and/or measured on MARS-5 L/N ≤35 at the first visit (corresponding to less than 80%). If the patient does not have asthma, it is MARS-5N ≤ 19
* If asthma: ACQ ≥1.2 or ACT ≤ 17 (partly uncontrolled asthma)
* SNOT-22 score ≥35 (partly uncontrolled CRS)
* Participation in the cross-sectional study at the initial visit to the Respiratory Clinic

Exclusion criteria:

Adherence:

* Foster score >80% and/or on MARS-5-L/N >35 points at the first visit
* Cannot read or speak Danish
* Severe psychiatric comorbidities
* Patients who have never taken systemic steroids
* After investigators' experience, will not be able to participate or comply with local treatment
* Does not give permission to look up data in FMK-online.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients referred to the Respiratory Clinic, ENT, RH, for evaluation of CRS/CRSwNP/CRSnNP and with or without asthma for biological treatment. They are classified according to the type of inflammation they have (type-2 or non-type-2), whether they have CRSwNP or CRSsNP, their adherence, comorbidity with asthma, and finally the severity of the disease. All patients are given standard questionnaires to assess CRS/CRSwNP/CRSnNP and asthma (STARR-15, SNOT22, ACQ, ACT, MARS-5-L/N, Fosterscore - routine questionnaires for all patients in the Respiratory Clinic).
  Patients for the project are recruited at the initial visit to the Respiratory Clinic. A nurse from the Respiratory Clinic will inform about the project and ask if the patient is interested in participating. If the patient is interested, a meeting will be arranged with a researcher from the research group (see section on information).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
P kortisol | 4 month follow-up
  Changes in P-cortisol i bloodsample

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Otorhinolaryngology, Head and Neck Surgery & Audiology, Copenhagen, Denamrk, Denmark

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/19/NCT05843019/Prot_ICF_000.pdf